CLINICAL TRIAL: NCT04788537
Title: Services to Enhance Social Functioning in Adults With Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 820694
Record Dates: First submitted 2021-03-02; First posted 2021-03-09 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Autism; Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome; Pervasive Developmental Disorder
Keywords: Autism; Autism Spectrum Disorder; Cognitive Behavioral Therapy
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Asperger Syndrome; Child Development Disorders, Pervasive | interventions — Drug Interactions

STUDY DESIGN:
Intervention Model Description: Participants randomly assigned to either the intervention group (50%) or nonintervention group (50%).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: Training to Understand and Navigate Emotions and Interactions (TUNE In)
- Nonintervention Group (No Intervention)

INTERVENTIONS:
Behavioral: Training to Understand and Navigate Emotions and Interactions (TUNE In) — A three-part cognitive behavioral treatment strategy to improve social functioning in adults with autism spectrum disorder. TUNE In includes components to address the many behavioral domains involved in social functioning, including social motivation, social anxiety, social cognition, social skills, and generalization of the skills to community settings.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to test a novel, three-part cognitive behavioral treatment strategy to improve social functioning in adults with autism spectrum disorder.

The treatment, named TUNE In (Training to Understand and Navigate Emotions and Interactions), includes components to address the many behavioral domains involved in social functioning, including social motivation, social anxiety, social cognition, social skills, and generalization of the skills to community settings.

The Investigators will test the efficacy of TUNE In to improve social functioning in adults with autism spectrum disorder (ASD), using a randomized controlled trial using the SRS-2 as the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of autism spectrum disorder

Exclusion Criteria:

* intellectual disability
* severe mood or psychotic symptoms experienced in the past 4 weeks
* severe self-injurious or aggressive behavior
* severe extrapyramidal motor or sedating side effects of medications
* concomitant participation in another social skills treatment program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Perelman School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be available through NIH NDAR registry
Time Frame: Deidentified data will be uploaded to NDAR upon completion of the trial

RESULTS

PARTICIPANT FLOW:
Groups:
- Nonintervention Group: Treatment As Usual
Period: Overall Study
Arm/Group | Intervention Group | Nonintervention Group
Started | 22 | 22
Completed | 18 | 20
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Nonintervention Group | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.82 (10.40) | 27 (8.76) | 27.91 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 21 | 21 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 17 | 19 | 36
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44
Shipley-2 - Vocabulary [Mean (Standard Deviation); unit: Scores on a Scale] — Scores on a scale of 100 = "Average" Vocabulary. Greater scores reflect greater verbal ability. Participants were required to score about 70 to qualify for study. The range of the scale has a minimum of 40 and a maximum of 140.
  Scores on a Scale | 118.77 (6.44) | 114.33 (12.23) | 117.16 (8.68)

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Social Responsiveness Scale, Second Edition (SRS-2) - Adult (Relative/Other Report)
Description: Scale ranges from 30 to 90 with higher T-scores indicating greater severity of autism symptomatology.
Time Frame: Baseline and Post-Treatment (~1 year after baseline)
Population: 2 Participants began but failed to complete TUNE In. 2 TAU participants lost to follow-up
Measure: Mean (Standard Deviation); unit: Scaled Score
Arm/Group | Intervention Group | Nonintervention Group
Number analyzed (Participants) | 20 | 22
Scaled Score
  Baseline | 68.67 (5.33) | 70.41 (6.70)
  Post-Treatment: number analyzed (Participants) | 18 | 20
  Post-Treatment | 66.08 (10.90) | 72.33 (6.04)
Statistical Analysis 1: Comparison: Intervention Group vs Nonintervention Group; Test type: Superiority — Linear mixed model regression; p = .006, Mixed Models Analysis; Slope = -1.58 — Slope reported is for Time x Group Interaction

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention Group | Nonintervention Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT04788537/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT04788537/SAP_001.pdf